CLINICAL TRIAL: NCT00373776
Title: Miltefosine for Mucosal Leishmaniasis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AB Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04--01
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2006-09-08 (Estimated); Status verified 2006-09

CONDITIONS: Leishmaniasis
Keywords: mucosal; leishmaniasis; miltefosine
MeSH Terms: conditions — Leishmaniasis | interventions — miltefosine

INTERVENTIONS:
Drug: miltefosine 2.5 mg/kg/day for 28 days

SUMMARY:
This trial will study miltefosine as a treatment for mucosal leishmaniasis.

DETAILED DESCRIPTION:
Treat bolivian mucosal leishmaniasis with miltefosine.

ELIGIBILITY:
Inclusion Criteria:

* Mucosal leishmaniasis

Exclusion Criteria:

* Abnormal liver function tests (LFT)
* Abnormal kidney function test
* Concomitant diseases

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2004-04; Study Completion 2006-05

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Jaime soto, MD, Principal Investigator — CIBIC
Locations (1):
- Palos Blancos, Bolivia